CLINICAL TRIAL: NCT06900829
Title: #AWARE.HIV Europe: Supporting Healthcare Professionals to Find Undiagnosed HIV in European Hospitals: An Effectiveness-implementation Trial.
Acronym: #aware hiv
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Casper Rokx (Other)
Collaborators: ViiV Healthcare (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Casper Rokx, Internist-infectiologist, Associate professor, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: MEC-2024-0236
Record Dates: First submitted 2025-02-24; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: HIV Infection; HIV; Stigma; Education; Prevention of Infection With HIV-1; Electronic Health Records
Keywords: hiv; stigma; linkage to care; linkage to prevention; electronic prompts; behavioural intervention; ICD-10 code based; audit and feedback
MeSH Terms: conditions — HIV Infections; Social Stigma; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Stepped wedge design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hiv team implemented (Experimental): A local hiv team will be implemented in a certain hospital. This will result in different activities, with a focus on:
  * audit and feedback (reminding health care professionals to test for hiv)
  * stigma reduction (raising awareness on existing hiv stigma towards hiv)
  * education (increasing knowledge on hiv among health care professionals)
  * linkage to prevention and care (improving pathways for hiv care and prevention)
  Interventions: Behavioral: HIV team implementation

INTERVENTIONS:
Behavioral: HIV team implementation — A local hiv team will be implemented in a certain hospital. This will result in different activities, with a focus on:
  * audit and feedback (reminding health care professionals to test for hiv)
  * stigma reduction (raising awareness on existing hiv stigma towards hiv)
  * education (increasing knowledge on hiv among health care professionals)
  * linkage to prevention and care (improving pathways for hiv care and prevention)

SUMMARY:
The #aware.hiv Europe study is a real-world, multicenter, stepped-wedge cluster randomized, effectiveness-implementation trial designed to evaluate whether the introduction of dedicated HIV teams in hospitals can improve HIV testing rates among patients presenting with HIV indicator conditions across ten European countries.

Study Design:

The study employs a stepped-wedge design, whereby clusters of hospitals transition sequentially from a control phase (routine care) to an intervention phase. All patient data are collected retrospectively from routine care, while prospective data are gathered at the healthcare professional level. The project spans four years and involves hospitals from the Netherlands, Belgium, United Kingdom, Germany, Spain, France, Italy, Romania, Poland, and Ukraine. This design allows for comparison of HIV testing rates and related outcomes before and after the implementation across different settings and time points.

Intervention:

The core intervention involves the establishment of hospital-based HIV teams. Each team is led by an HIV specialist and supported by nurses and data collectors. Their responsibilities include:

Identification and Surveillance: Screening routine electronic health records for HIV indicator conditions using predefined ICD-10 codes and verifying cases that warrant HIV testing.

Audit & Feedback: Providing targeted recommendations to treating physicians when an HIV test is indicated but has not been performed, thereby prompting action.

Education & Training: Delivering training sessions to healthcare professionals to improve their knowledge and attitudes towards HIV testing, prevention, and care.

Enabling Environment: Implementing digital solutions and other support mechanisms to streamline testing processes, reduce stigma, and enhance overall guideline adherence.

Linkage to prevention: Improving linkage to the locally available preventive services.

The intervention is intended to integrate seamlessly into routine hospital care, thereby reinforcing existing guidelines while addressing the current diagnostic testing gap.

Endpoints and Outcome Measures:

Primary Endpoint:

The change in HIV testing rate among patients diagnosed with HIV indicator conditions before and after the implementation of HIV teams.

Key Secondary Endpoints:

The change in the incidence of new HIV diagnoses among patients with HIV indicator conditions.

Variations in HIV testing rates across different countries, medical specialties, and types of indicator conditions, as well as over time.

Assessment of the cascade of HIV diagnosis, including the proportion of patients identified with an indicator condition, the offer and acceptance of HIV testing, and documented reasons for non-testing.

Evaluation of the cascade of HIV care and prevention, including linkage to HIV care, achievement of viral suppression, and referral and uptake of preventive services.

Changes in healthcare professionals' knowledge, attitudes, and levels of stigma towards HIV.

Implementation outcomes such as fidelity of HIV team activities, resource utilization, cost-effectiveness, and sustainability of the intervention.

Analysis of contextual factors, barriers, and facilitators impacting the implementation process, using established frameworks like CFIR and RE-AIM.

Impact:

By introducing HIV teams and systematically monitoring their effect on HIV testing practices, the study aims to enhance early HIV diagnosis and improve patient outcomes. The findings will contribute to evidence-based guidelines and may promote the adoption of similar interventions across European healthcare settings, ultimately reducing HIV-associated morbidity, mortality, and transmission rates.

This project not only addresses a critical diagnostic gap in HIV care but also provides valuable insights into the effective implementation of complex interventions in routine clinical practice.

ELIGIBILITY:
Since this study involves screening individuals presenting to a specific hospital through a hospital-wide intervention, the inclusion and exclusion criteria are established at the hospital level.

Inclusion Criteria:

1. Standard of care: HIV testing for HIV indicator conditions should be part of routine care in the country, and any prevailing guidelines on HIV testing and prevention policies can be integrated.
2. Management approval: Hospital management must be willing to allocate resources and provide authorization for the proposed activities, including Surveillance, Audit & Feedback, Education & Training, Linkage to Prevention, and fostering an Enabling Environment, including stigma reduction.
3. Resources: Assembling an HIV team led by a local HIV expert should be viable considering the available human resources.
4. Data collection: There should be an IT specialist and IT infrastructure capable of flagging a pre-defined set of HIV indicator conditions and monitoring the project's implementation effects with feedback loops to healthcare professionals.
5. Quality assurance: Continuous linkage for care and access to antiretroviral therapy must be assured.
6. Ethics and Regulatory Compliance: Provision for ethical and regulatory compliance is necessary.

Exclusion Criteria:

Any hospital that does not meet the inclusion criteria will be excluded from participation. We will not use data of patients who have objected against the use of their data for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5200 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
HIV testing rate in patients with HIV indicator conditions | Comparison between 1 year of implementation and a control phase lasting between 6 to 18 months, depending on the site's randomization in the stepped-wedge trial design.
  Proportion of patients diagnosed with an HIV indicator condition who receive an HIV test, compared between the control and implementation phases.

SECONDARY OUTCOMES:
HIV incidence in patients with HIV indicator conditions | Comparison between 1 year of implementation and a control phase lasting between 6 to 18 months, depending on the site's randomization in the stepped-wedge trial design.
  Number of newly diagnosed HIV infections among patients with an HIV indicator condition, compared between the control and implementation phases.
Subgroup analysis 1: HIV testing rate by country and region | Comparison between 1 year of implementation and a control phase lasting between 6 to 18 months, depending on the site's randomization in the stepped-wedge trial design.
  Difference in HIV testing rate within and between countries, as well as between geographic regions (West: Netherlands, Belgium, UK, Germany; South: France, Italy, Spain; East: Poland, Romania, Ukraine), comparing the control and implementation phases.
Subgroup analysis 2: HIV testing rate by HIV indicator condition | Comparison between 1 year of implementation and a control phase lasting between 6 to 18 months, depending on the site's randomization in the stepped-wedge trial design.
  Difference in HIV testing rate across different HIV indicator conditions, comparing the control and implementation phases.
Subgroup analysis 3: HIV testing rate by medical specialty | Comparison between 1 year of implementation and a control phase lasting between 6 to 18 months, depending on the site's randomization in the stepped-wedge trial design.
  Difference in HIV testing rate across medical specialties, comparing the control and implementation phases.
Subgroup analysis 4: HIV testing rate over time | Comparison between 1 year of implementation and a control phase lasting between 6 to 18 months, depending on the site's randomization in the stepped-wedge trial design.
  Change in HIV testing rate over time, comparing the control and implementation phases.
Cascade 1: The cascade of HIV diagnosis | Comparison between 1 year of implementation and a control phase lasting between 6 to 18 months, depending on the site's randomization in the stepped-wedge trial design.
  Proportion of patients with a confirmed HIV indicator condition (focus population) who were offered an HIV test (reach) and who accepted testing (uptake), compared between the control and implementation phases.
Cascade 1b: The cascade of HIV diagnosis - reasons for not testing for HIV | Comparison between 1 year of implementation and a control phase lasting between 6 to 18 months, depending on the site's randomization in the stepped-wedge trial design.
  Qualitative analysis of documented reasons why patients with an HIV indicator condition did not receive an HIV test. Reasons will be classified according to predefined categories used in the study database:
  No reason registered (1) Patient was not seen again (2) Advice to the general practitioner or public health to test (3) No perceived indication or risk factors (4) Alternative diagnosis/explanation (5) No recommendation in local protocol (6) Patient refused (7) Shared decision-making not to test (8) Lack of time or opportunity (9) Planned but not performed (10) Already tested (confirmed) (11) Already tested (not confirmed or inadequate according to the SOP) (12) Palliative care or patient deceased during follow-up (13) Other (14)
Cascade 1c: The cascade of HIV diagnosis - descriptions of existing consent procedures in different hospital sites | Description of consent procedures as documented during the 1-year implementation phase across different hospital sites.
  Qualitative description of the consent procedures in place for HIV testing across different hospital sites. This includes:
  The types of consent procedures in use, such as verbal or written consent. National or institutional guidelines or local standard procedures that shape consent practices.
  Data will be collected per site to document existing practices without assessing implementation or adherence.
Cascade 2: The cascade of HIV care | Comparison between 1 year of implementation and a control phase lasting between 6 to 18 months, depending on the site's randomization in the stepped-wedge trial design.
  Proportion of patients with a confirmed HIV indicator condition who were newly diagnosed with HIV (focus population) and subsequently linked or re-linked to routine HIV care (reach), with viral suppression as an indicator of successful engagement in care (uptake), compared between the control and implementation phases.
Cascade 3: The cascade of HIV prevention | Comparison between 1 year of implementation and a control phase lasting between 6 to 18 months, depending on the site's randomization in the stepped-wedge trial design.
  Proportion of patients with a confirmed HIV indicator condition who met the eligibility criteria for HIV prevention (focus population), were appropriately referred to prevention services (reach), and engaged in prevention interventions (uptake), compared between the control and implementation phases.
HIV stigma indicators among health care professionals | Assessed at baseline (before implementation) and at 12 months (after 1 year of implementation).
  Descriptive assessment of self-reported HIV stigma among licensed healthcare professionals, including physicians, nurse practitioners, and physician assistants, before and after implementation. Stigma will be measured using a validated questionnaire developed by the Health Policy Project and USAID, and adapted from the ECDC survey published in Annex 1 of the report: "HIV stigma in the healthcare setting. Monitoring implementation of the Dublin Declaration on partnership to fight HIV/AIDS in Europe and Central Asia 2024."
  The survey includes self-reported responses on multiple dimensions of HIV stigma, expressed as percentages of participants reporting:
  1. Fear of HIV infection
  2. Institutional facilitators and barriers
  3. Negative attitudes towards people with HIV
  4. Observed stigma in clinical settings.
  This is a descriptive outcome measure, reporting the proportion of participants endorsing each stigma-related item before and after the intervention.
Implementation science 1: Assessment of key barriers and facilitators over time (CFIR) | Every 3 months during the implementation phase (first year). Every 6 months during the continuation phase (up to 3 years post-implementation).
  Description:
  Descriptive assessment of perceived barriers and facilitators to implementing and sustaining the HIV team intervention in hospital settings. Barriers and facilitators will be assessed based on a structured survey, capturing key constructs from the Consolidated Framework for Implementation Research (CFIR): Intervention characteristics, Outer setting, Inner setting, Characteristics of individuals and the Implementation process.
  Survey items will be derived from a systematic review of barriers and facilitators to HIV indicator condition-based testing. The review will be published separately.
  Data will be collected via an online survey in Castor, administered to the HIV team lead at each participating site
Implementation science 2: Reach: Proportion of patients benefiting from HIV team-supported testing | Measured during the implementation phase (1st year) and continuation phase (2nd year), compared to the control phase (6-18 months before implementation).
  Proportion of patients with HIV indicator conditions who received an HIV test with direct (= feedback) or indirect (= other implementation strategies) involvement of the HIV team, stratified by:
  * Country, hospital, and specialty to assess variation in reach
  * Equity analysis: evaluating differences in testing uptake by age and sex
Implementation science 3a: Effectiveness: Impact on HIV diagnosis rate | Measured during the implementation phase (1st year) and continuation phase (2nd year), compared to the control phase (6-18 months before implementation).
  Proportion of individuals who test HIV-positive among:
  All individuals tested for HIV (primary analysis). All individuals identified with an HIV indicator condition (secondary analysis).
Implementation science 3b: Effectiveness: Impact on disease stage at presentation | Measured during the implementation phase (1st year) and continuation phase (2nd year), compared to the control phase (6-18 months before implementation).
  Assessment of the impact of the HIV indicator condition-based testing approach on CD4 count at HIV diagnosis, measured as a continuous variable to assess shifts in stage at presentation.
  Primary analysis:
  Mean CD4 count at HIV diagnosis in the intervention phase vs. control phase (continuous variable).
  Secondary analysis:
  Distribution of CD4 counts at diagnosis (percentiles and quartiles) to evaluate changes in the proportion of late-stage diagnoses.
  Proportion of patients diagnosed with advanced HIV (CD4 <200 cells/µL) in both phases.
  Proportion of patients diagnosed with late-stage HIV (CD4 <350 cells/µL) in both phases.
  Proportion of patients diagnosed at higher CD4 thresholds (e.g., >500 cells/µL) to assess shifts towards earlier diagnosis.
Implementation science 4a: Adoption of HIV Indicator Condition-based testing | Measured during the implementation phase (1st year) and continuation phase (2nd year), compared to the control phase (6-18 months before implementation).
  Hospital adoption rate (%): Proportion of participating hospitals that have adopted all core components of HIV indicator condition-based testing.
  as well as: Degree of adoption across the hospital (%): Proportion of hospital departments (inpatients, outpatients, SEH, IC) that are included in the surveillance of HIV indicator condition-based testing.
Implementation science 5a: Implementation - Fidelity to the implementation strategies | Measured during the implementation phase (1st year) and continuation phase (2nd year)
  This outcome assesses the degree to which the #aware.hiv Europe implementation strategies were delivered as intended across participating hospitals.
  Percentage of flagged potential HIV indicator conditions that were assessed by the HIV team (surveillance) Percentage of untested indicator conditions for which HIV testing advice was provided to physicians (feedback) Number of teaching sessions delivered compared to the intended frequency, with a minimum of one session every three months in the implementation phase (teaching).
  Number of stigma-reducing events organized, with a minimum requirement of one event in the implementation phase (stigma).
Implementation science 5b: Implementation - Adaptation of the implementation strategies | This will be assessed every three months during the implementation phase, and every 6 months in the first year of the continuation phase..
  This outcome assesses the extent to which the #aware.hiv Europe implementation strategies were adapted to fit the local context while maintaining core components across participating hospitals.
  The number and type of modifications made to the implementation strategy at the hospital level will be assessed using qualitative data collected via a structured questionnaire. Responses will be categorized according to the key components of the implementation strategy:
  * Audit and Feedback
  * Teaching and Education
  * Enabling Environment (including stigma reduction)
  * Linkage to Prevention
Implementation science 5c: Implementation - Acceptability and appropriateness of the implementation strategies | As part of the stigma questionnaire before and after the implementation phase.
  This outcome assesses how acceptable and appropriate the #aware.hiv Europe implementation strategies are perceived by healthcare professionals authorised to request HIV tests, using questions embedded in the hospital-wide stigma questionnaire.
Cost-effectiveness | The one-year implementation phase will be compared to the preceding control phase, and the continuation phase (second year) will be compared to both the implementation and control phases to assess cost-effectiveness.
  Cost-effectiveness will be estimated by calculating the budget impact and Quality-Adjusted Life Years (QALYs) saved to define an Incremental Cost-Effectiveness Ratio (ICER).
Epidemiological impact | The one-year implementation phase will be compared to the control phase, and the continuation phase (second year) will be compared to both preceding phases.
  The epidemiological impact will be estimated by quantifying the number of earlier HIV diagnoses achieved through the intervention, and modelling the resulting reduction in the number of person-years spent living with undiagnosed HIV. In addition, the number of secondary HIV infections potentially averted due to earlier diagnosis and treatment initiation will be estimated.
  Estimate the reduction in average time from infection to diagnosis based on clinical data and literature.
  Calculate the total number of person-years with undiagnosed HIV prevented through earlier detection.
  Use published transmission rates for undiagnosed individuals to model the number of secondary infections averted.
  If available, incorporate local or national modelling tools (e.g., ECDC HIV Modelling Tool) to support these estimates.

CONTACTS AND LOCATIONS:
Overall Officials: Casper Rokx, Infectiologist, associate prof, Principal Investigator — Erasmus Medical Center

IPD SHARING:
Plan to Share IPD: No
While aggregated results may be published, the protocol does not support the sharing of individual-level data.

REFERENCES:
- [Background] Jordans CCE, Vliegenthart-Jongbloed K, Osbak KK, Hanssen JLJ, van Beek J, Vriesde M, van Holten N, Dorama W, van der Sluis D, de Steenwinkel J, van Kampen J, Verbon A, Roukens AHE, Rokx C. Implementing HIV teams sustainably improves HIV indicator condition testing rates in hospitals in the Netherlands: the #aware.hiv clinical trial. AIDS. 2025 Jul 1;39(8):995-1004. doi: 10.1097/QAD.0000000000004167. Epub 2025 Mar 18. PMID 40053486
- [Background] Jordans CCE, Vliegenthart-Jongbloed KJ, van Bruggen AW, van Holten N, van Beek JEA, Vriesde M, van der Sluis D, Verbon A, Roukens AHE, Stutterheim SE, Rokx C. Unmasking Individual and Institutional HIV Stigma in Hospitals: Perspectives of Dutch Healthcare Providers. AIDS Behav. 2024 Sep;28(9):3184-3195. doi: 10.1007/s10461-024-04404-0. Epub 2024 Jun 13. PMID 38869755
- [Background] Vliegenthart-Jongbloed KJ, Vasylyev M, Jordans CCE, Bernardino JI, Nozza S, Psomas CK, Voit F, Barber TJ, Skrzat-Klapaczynska A, Sandulescu O, Rokx C; #aware.hiv Europe Project. Systematic Review: Strategies for Improving HIV Testing and Detection Rates in European Hospitals. Microorganisms. 2024 Jan 25;12(2):254. doi: 10.3390/microorganisms12020254. PMID 38399659
- See also: Related Info — https://awarehiv.com/